CLINICAL TRIAL: NCT01782261
Title: Pilot Study on Incretin Effect on the Immunological Phenotype in Healthy Subjects and in Type 1 Diabetic Subjects
Brief Title: Incretin Effect on the Immunological Phenotype
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADPP004; 2011-006300-12 (EudraCT Number)
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes
Keywords: autoimmune disease; diabetes type 1; incretin effect
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases | interventions — Liraglutide; saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): Liraglutide subcutaneous injection every day. first week 0.6mg, week 2-4 1.2mg.
  Interventions: Drug: Liraglutide
- Saxagliptin (Active Comparator): Saxagliptin 5mg tablet by mouth every day for 4 weeks
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Liraglutide — once daily subcutaneous injection
  Other Names: Victoza
  Arms: Liraglutide
Drug: Saxagliptin — once daily tablet
  Other Names: Onglyza
  Arms: Saxagliptin

SUMMARY:
Assessment of the effect of incretin based therapies (Liraglutide and Saxagliptin) on immune cells in healthy subjects and patients with type 1 diabetes

DETAILED DESCRIPTION:
Assessment of immunological effects of Saxagliptin and Liraglutide on immune cells of the peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

-healthy subjects or patients with type 1 diabetes

Exclusion Criteria:

* pregnancy
* treatment with GLP-1-Analoga (Liraglutide, Exenatide)
* treatment with DPP4-inhibitor (Sitagliptin, Vildagliptin, Saxagliptin)
* chronic disease including a long-term medication over 4 weeks per year (except type 1 diabetes)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Increase of regulatory FOXP3+ T cells | 4 weeks
  the effects of incretin based therapy on regulatory FOXP3+ T cells will be measured at baseline and after 4 weeks

SECONDARY OUTCOMES:
Immunophenotyping | 4 weeks
  The effect of incretin based therapy on circulating immune cells and cytokine secretion at baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, Professor, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No